CLINICAL TRIAL: NCT01414114
Title: A Single-arm, Open-label, Multicenter, Dose Titration Study of KAI-4169 to Treat Secondary Hyperparathyroidism in Hemodialysis Subjects With Chronic Kidney Disease-Mineral and Bone Disorder
Brief Title: Etelcalcetide to Treat Secondary Hyperparathyroidism in Hemodialysis Patients With Chronic Kidney Disease-Mineral and Bone Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KAI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAI-4169-005; 20120331 (Other: Amgen, Inc)
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Clinical Trial, Phase 2; Renal Dialysis; Secondary Hyperparathyroidism; Chronic kidney disease-mineral and bone disorder; Parathyroid hormone
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etelcalcetide (Experimental): Participants received etelcalcetide three times a week (TIW) administered by intravenous bolus injection at the end of each hemodialysis session for 12 weeks. The starting dose was 5 mg and may have been titrated every 4 weeks based on the preceding serum parathyroid hormone (PTH) and corrected calcium (cCa) levels to a maximum dose of 20 mg per hemodialysis session in order to achieve the targeted PTH range while maintaining serum calcium within an acceptable range.
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — Administered 3 times a week by bolus injection into the venous line of the dialysis circuit after the end of hemodialysis.
  Other Names: KAI-4169; AMG 416; Parsabiv™

SUMMARY:
The purpose of this study is to evaluate the effect of thrice weekly intravenous (IV) administration of etelcalcetide in the treatment of secondary hyperparathyroidism (SHPT) in hemodialysis patients with chronic kidney disease-mineral and bone disorder (CKD-MBD).

ELIGIBILITY:
Inclusion Criteria:

* Subjects provides written informed consent
* Screening intact PTH (iPTH) ≥ 350 pg/mL and corrected calcium ≥ 8.5 mg/dL
* Hemoglobin ≥ 8.5 g/dL
* Serum transaminases (alanine transaminase [ALT], aspartate transaminase [AST]) less than 2.5 times the upper limit of normal
* Adequate hemodialysis three times per week

Exclusion Criteria:

* History or symptomatic ventricular dysrhythmias
* History of angina pectoris or congestive heart failure
* History of myocardial infarction, coronary angioplasty, or coronary artery bypass grafting within the past 6 months
* History of or treatment for seizure disorder within the last 12 months
* Postdialysis systolic blood pressure > 180 mmHg or diastolic blood pressure > 90 mmHg
* Serum magnesium below the lower limit of normal at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-12-05; Primary Completion 2012-05-21 (Actual); Study Completion 2012-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Bell, MD, Study Director — KAI Pharmaceuticals

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 centers in the United States from 05 December 2011 (first participant enrolled) to 21 May 2012 (last participant completed follow-up).
Period: Overall Study
Arm/Group | Etelcalcetide
Started | 37
Completed | 32 (Completed 12-week treatment period)
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (13.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 19
Race [Count of Participants; unit: Participants]
  White | 18
  Black or African American | 19
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 26
Parathyroid Hormone (PTH) [Mean (Standard Deviation); unit: pg/mL] | 853.4 (644.25)
Parathyroid Hormone Category [Count of Participants; unit: Participants]
  ≤ 700 pg/mL | 22
  > 700 pg/mL | 15
Corrected Calcium [Mean (Standard Deviation); unit: mg/dL] | 10.1 (0.62)
Phosphorus [Mean (Standard Deviation); unit: mg/dL] | 5.7 (1.38)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Parathyroid Hormone (PTH) During the Efficacy Period
Description: Baseline was defined as the average of 3 predialysis PTH results obtained within 3 weeks of and prior to the first dose of study drug. The efficacy period (defined as the period from 14 days prior to and 3 days after the last dose of study drug) value was the mean of the prehemodialysis values obtained during that period.
Time Frame: Baseline and the efficacy period, defined as from 14 days prior to and 3 days after the last dose of study drug (approximately days 68 - 85 for participants who completed 12 weeks of treatment)
Population: The modified intent-to-treat population (all participants who were randomized and received treatment) with available data at both time points.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Baseline PTH ≤ 700 pg/mL: Participants with baseline PTH ≤ 700 pg/mL
- Baseline PTH > 700 pg/mL: Participants with baseline PTH > 700 pg/mL
Arm/Group | Etelcalcetide | Baseline PTH ≤ 700 pg/mL | Baseline PTH > 700 pg/mL
Number analyzed (Participants) | 36 | 21 | 15
percent change | -53.6 (21.42) | -55.6 (19.65) | -50.8 (24.12)

2. Secondary Outcome: Percentage of Participants With ≥ 30% Reduction in PTH From Baseline During the Efficacy Period
Description: The efficacy period (defined as the period from 14 days prior to and 3 days after the last dose of study drug) value was the mean of the prehemodialysis values obtained during that period.
Time Frame: as for outcome 1
Population: Modified intent-to-treat population with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etelcalcetide | Baseline PTH ≤ 700 pg/mL | Baseline PTH > 700 pg/mL
Number analyzed (Participants) | 36 | 21 | 15
percentage of participants | 89 [73.9 to 96.9] | 95 [76.2 to 99.9] | 80 [51.9 to 95.7]

3. Secondary Outcome: Percentage of Participants With PTH ≤ 300 pg/mL During the Efficacy Period
Description: as for outcome 2
Time Frame: The efficacy period, defined as from 14 days prior to and 3 days after the last dose of study drug (approximately days 68 - 85 for participants who completed 12 weeks of treatment)
Population: Modified intent-to-treat population with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etelcalcetide | Baseline PTH ≤ 700 pg/mL | Baseline PTH > 700 pg/mL
Number analyzed (Participants) | 36 | 21 | 15
percentage of participants | 56 [38.1 to 72.1] | 76 [52.8 to 91.8] | 27 [7.8 to 55.1]

4. Secondary Outcome: Percent Change From Baseline in Corrected Calcium During the Efficacy Period
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Modified intent-to-treat population with available data at both time points
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etelcalcetide | Baseline PTH ≤ 700 pg/mL | Baseline PTH > 700 pg/mL
Number analyzed (Participants) | 36 | 21 | 15
percent change | -15.1 (5.76) | -13.0 (4.83) | -17.9 (5.91)

5. Secondary Outcome: Percent Change From Baseline in Phosphorus During the Efficacy Period
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Modified intent-to-treat population with available data at both time points
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etelcalcetide | Baseline PTH ≤ 700 pg/mL | Baseline PTH > 700 pg/mL
Number analyzed (Participants) | 36 | 21 | 15
percent change | -10.4 (19.78) | -7.7 (21.92) | -14.2 (16.27)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 4 weeks after the last dose; 16 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Etelcalcetide
Serious Adverse Events (participants affected / at risk) | 3/37
Other Adverse Events (participants affected / at risk) | 18/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etelcalcetide (N=37)
Acute myocardial infarction (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etelcalcetide (N=37)
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Blood calcium decreased (Investigations) | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.